CLINICAL TRIAL: NCT02747810
Title: Pilot Study: Foot Neuromodulation for Nocturnal Enuresis in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We have decided not to test the newly designed TENS device
Sponsor: Heidi Stephany (Other)
Collaborators: CMI's Early-Stage Medical Technology Research and Development 2015 PILOT FUNDING PROGRAM (Unknown)
Responsible Party: Sponsor-Investigator, Heidi Stephany, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15070130
Record Dates: First submitted 2016-04-05; First posted 2016-04-22 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Bedwetting
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- New TENS design (Experimental): To determine the function and safety of the strap design by evaluating the electrical connection to electrode, 2) the security in the insole and the electronic unit, and 3) facilitating observation and hand access to the top panel for adjusting the stimulation strength. 4) to elicit toe twitching with stimulation of tribal nerve
  Interventions: Device: NewTENS Design

INTERVENTIONS:
Device: NewTENS Design — This device functions the same as the FDA approved TENS unit, but provides a small, inexpensive unit that will be easy for a child to use. The stimulation characteristics include a continuous frequency of 5 Hz, pulsewidth 0.2 ms, and intensity 2-4 times the threshold voltage required for inducing toe twitching - or the intensity that the subject feels comfortable with. The subjects will also be instructed how to use the stimulator and where to attach the electrodes on the foot at the beginning of the study. The investigator will provide the stimulator and electrodes. The subjects will be asked to wear socks to prevent the electrodes from detachment and to stop the stimulation during walking or in any non-resting situation. Subjects will be asked to use the stimulator for a MINIMUM of 60 minutes in the evening prior to bedtime at home for two weeks. They will be encouraged to use the stimulator for more time than the minimum as long as they accurately record the total duration.

SUMMARY:
Background: Previous animal model studies at the University of Pittsburgh have shown a significant impact on inhibiting bladder over activity and increasing bladder capacity with neuromodulation techniques, specifically tibial nerve stimulation. This has been translated into adult clinical trials through the department of urology. Through the use of a commercially available subcutaneous nerve stimulator placed on the dorsum of the foot, researchers were able to demonstrate a significant increase in bladder capacity and the delay of voiding sensation for up to 5 hours after stimulation in eight healthy subjects. This prompted the clinical trial approved under IRB PRO13020474 which is currently enrolling patients.

The incidence of night-time overactive bladder leading to nocturnal enuresis (bed wetting) is very common in the pediatric and teenage population, particularly in patients without daytime bladder over activity symptoms. When behavioral modification (i.e. refraining from night-time fluid consumption and bladder irritants, and bed wetting alarms for timed voiding) fails which it often does there is a paucity of effective and safe treatment options. Medications can be tried, but generally these are from the tricyclic antidepressant family and carry significant side effects limiting the use.

Aim: Researchers aim to utilize the same technology currently being studied under IRB PRO14080250. Electrical stimulation will be applied to the foot via skin surface electrodes for a minimum of 1 hour before bed for 2 weeks to 5 normal subjects. Normal Subjects will be asked to complete a questionnaire about any skin irritation or experiences of toe twitching while wearing the newly designed TENS device, during a return visit with Dr. Stephany. The primary outcomes of this study are safety and functionality of the New TENS unit

DETAILED DESCRIPTION:
Nocturnal Enuresis is a very common and difficult to treat problem in the pediatric population which can have significant negative impact on a child's quality of life. Apart from medications which can have significant side effects limiting the use, there is a lack of effective and safe treatment options for children with frequent nocturnal enuresis. If foot stimulation prior to bed does indeed improve the frequency of nocturnal enuresis, it may provide a safe and non-invasive therapeutic option.

To achieve the aims Dr. Tai will work closely with Dr. Sun and Dr. Jia to design and develop a small, inexpensive, and easy-to-use stimulator for foot neuromodulation, and test its safety and usability in 5 healthy subjects for a 2-week period. . The straps in the design have three functions: 1) making an electrical connection to electrode, 2) securing the insole and the electronic unit, and 3) facilitating observation and hand access to the top panel for adjusting the stimulation strength.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 5 to 16 years old without any specific nocturnal enuresisneurological, disorder or urinary tract infection.
2. Currently having no daytime overactive bladder symptoms, i.e. urinary frequency, urgency, or daytime incontinence

Exclusion Criteria:

1. Patients with nocturnal enuresis and day time symptoms will be excluded from this study.
2. Children with known neurological disorders which may be contributing to nocturnal enuresis episodes
3. Children who are not adequately potty trained
4. Children with significant daytime symptoms of overactive bladder including frequency, urgency, and daytime incontinence
5. Children who do not tolerate initial stimulation training session in the urology clinic upon enrollment
6. Children with any implantable medical devices such as a pacemaker will be excluded from the study

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Questionnaire | 2 weeks
  Subjects will be asked to record the intensity at which they see the big toe twitching and where they keep the intensity over the hour of stimulation. They will also record if any issues with the unit or any side effects, such as pain or foot irritation. They will document the time of starting and finishing stimulation.

SECONDARY OUTCOMES:
Night Time log | 2 weeks
  Participants will complete a night time log to determine of the new design works at preventing night time wetting

CONTACTS AND LOCATIONS:
Overall Officials: Heidi A Stephany, MD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No